CLINICAL TRIAL: NCT02555020
Title: Effect of Preoperative Oral Carbohydrates on Quality of Recovery: Randomized Controlled Trial
Brief Title: Effect of Preoperative Oral Carbohydrates on Quality of Recovery
Acronym: laparoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Joon Seong Park, GangNam Severance Hospital, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 3-2015-0158
Record Dates: First submitted 2015-09-11; First posted 2015-09-21 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Evidence of Cholecystectomy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Allocated to MN NPO group, (Experimental): 1. Patients was administered in hospital
  2. Randomization
  3. Patient was allocated to MN group
  4. Patients were NPO from mid night (MN) to Surgery
  Interventions: Dietary Supplement: Allocated to MN NPO group,
- Allocated to Placebo group (Placebo Comparator): 1. Patients was administered in hospital
  2. Randomization
  3. Patient was allocated to Placebo group
  4. Patients received 400 mL of water 12 hours before anesthesia and 400 mL 2 hours before anesthesia.
  Interventions: Dietary Supplement: Allocated to Placebo group
- Allocated to Carbohydrated group (Active Comparator): 1. Patients was administered in hospital
  2. Randomization
  3. Patient was allocated to Carbohydrated group
  4. Patients received 400 mL of oral isotonic glucose (No NPO®, Daesang, Korea) 12 hours before anesthesia and 400 mL 2 hours before. CHL composition was standard: 12.5 g of carbohydrate per 100 mL, 12% monosaccharide, 12% disaccharide, 76% polysaccharide, 250 mOsm/kg and 50 kcal.
  Interventions: Dietary Supplement: Allocated to Carbohydrated group

INTERVENTIONS:
Dietary Supplement: Allocated to Carbohydrated group — Patients received 400 mL of oral isotonic glucose (No NPO®, Daesang, Korea) 12 hours before anesthesia and 400 mL 2 hours before. CHL composition was standard: 12.5 g of carbohydrate per 100 mL, 12% monosaccharide, 12% disaccharide, 76% polysaccharide, 250 mOsm/kg and 50 kcal.
  Arms: Allocated to Carbohydrated group
Dietary Supplement: Allocated to Placebo group — Patients received 400 mL of oral free water (Placebo) 12 hours before anesthesia and 400 mL 2 hours before.
  Arms: Allocated to Placebo group
Dietary Supplement: Allocated to MN NPO group, — Patients received NPO from MN.
  Arms: Allocated to MN NPO group,

SUMMARY:
Carbohydrate loading is an important component of enhanced recovery pathways. Preoperative carbohydrate treatments have been widely adopted as part of enhanced recovery after surgery (ERAS) or fast-track surgery protocols. Although fast-track surgery protocols have been widely investigated and have been shown to be associated with improved postoperative outcomes, some individual constituents of these protocols, including preoperative carbohydrate treatment, have not been subject to such robust analysis.To assess the effects of preoperative carbohydrate treatment, compared with placebo or preoperative fasting, on postoperative recovery and insulin resistance in adult patients undergoing elective surgery.

DETAILED DESCRIPTION:
Patients received 400 mL of oral isotonic glucose (No NPO®, Daesang, Korea) 12 hours before anesthesia and 400 mL 2 hours before. CHL composition was standard: 12.5 g of carbohydrate per 100 mL, 12% monosaccharide, 12% disaccharide, 76% polysaccharide, 250 mOsm/kg and 50 kcal.

ELIGIBILITY:
Inclusion Criteria:

1. ASA (I/II)
2. Laparoscopic cholecystectomy.
3. KAROFSKY PERFORMANCE SCALE >70,
4. No history of major operation

Exclusion Criteria:

1. DM patients
2. GE reflux Hx patients.
3. No- compliance,
4. Previous Abdominal Surgery History

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2016-12-23 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery score using the QoR-40 Questionnaire | We check the QoR-40 at POD1 after cholecystectomy , an expected average 3days
  We check the QoR-40 Questionnaire at discharge day

REFERENCES:
- [Derived] Lee JS, Song Y, Kim JY, Park JS, Yoon DS. Effects of Preoperative Oral Carbohydrates on Quality of Recovery in Laparoscopic Cholecystectomy: A Randomized, Double Blind, Placebo-Controlled Trial. World J Surg. 2018 Oct;42(10):3150-3157. doi: 10.1007/s00268-018-4717-4. PMID 29915988